CLINICAL TRIAL: NCT03108287
Title: Adding Bismuth to Rabeprazole-based First-line Triple Therapy Does Not Improve the Eradication of Helicobacter Pylori
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KMUH-IRB-20120028
Record Dates: First submitted 2017-03-23; First posted 2017-04-11 (Actual); Last update posted 2017-04-24 (Actual); Status verified 2017-03

CONDITIONS: Helicobacter Pylori Infection
MeSH Terms: interventions — Rabeprazole; Amoxicillin; Clarithromycin; bismuth tripotassium dicitrate

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- RAK therapy (Active Comparator): rabeprazole+amoxicillin+clarithromycin
  Interventions: Drug: RAK therapy
- RBAK therapy (Active Comparator): rabeprazole+amoxicillin+clarithromycin+bismuth subcitrate
  Interventions: Drug: RBAK therapy

INTERVENTIONS:
Drug: RAK therapy — rabeprazole 20mg, amoxicillin 1g and clarithromycin 500mg twice-daily
  Other Names: rabeprazole, amoxicillin, clarithromycin
  Arms: RAK therapy
Drug: RBAK therapy — rabeprazole 20mg, amoxicillin 1g and clarithromycin 500mg, bismuth subcitrate 360mg twice-daily
  Other Names: rabeprazole, amoxicillin, clarithromycin, bismuth subcitrate
  Arms: RBAK therapy

SUMMARY:
This randomized controlled study aimed to evaluate whether adding bismuth to the standard first-line triple therapy could improve the eradication rate of Helicobacter pylori (H. pylori). A total of 162 patients with H. pylori infection were randomly assigned to either the 7-day triple therapy group (n = 81) or the bismuth plus triple therapy group (n = 81). The triple therapy (RAK) contained the twice-daily dosage of rabeprazole 20mg, amoxicillin 1g and clarithromycin 500mg. In the RBAK group, bismuth subcitrate 360 mg twice daily was added to the RAK regimen.

DETAILED DESCRIPTION:
Once confirmed with H. pylori infection and having signed the informed consent, participants were randomly assigned to either the standard triple-therapy group (RAK: rabeprazole 20 mg, amoxicillin 1 g and clarithromycin 500 mg, all twice daily for 7 days) or the bismuth plus standard triple-therapy group (RBAK: rabeprazole 20 mg, bismuth subcitrate 360 mg, amoxicillin 1 g and clarithromycin 500 mg, all twice daily for 7 days). A computer-generated random number was chosen for randomization. The patients and physicians were not blinded to the therapy assigned.

After completion of H. pylori eradication therapy, participants were asked to come back for collection of the information on any adverse event of drug compliance. In order to avoid false negative results, they were also asked to have a 4-week proton pump inhibitor, antibiotic and bismuth washout period before further examination of H. pylori status. The second endoscopy with rapid urea test, histology and culture or 13 C-urea breath test (UBT) for those who refused endoscopic exams was carried out at the end of the washout period. Those who did not return to confirm their H. pylori status were deemed as treatment failure in intention-to-treat (ITT) analysis.

ELIGIBILITY:
Inclusion Criteria:

1. male or non-pregnant female aged more than 20 y/r
2. H.pylori-infected
3. mental and legal ability to give a written informed consent

Exclusion Criteria:

1. allergy to any drug in the study
2. prior gastric surgery, severe concomitant diseases (e.g., decompensate liver cirrhosis, uremia, gastric cancer)
3. previous H. pylori eradication therapy
4. pregnancy or lactation.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Actual)
Dates: Start 2013-04-01 (Actual); Primary Completion 2015-01-31 (Actual); Study Completion 2015-02-28 (Actual)

PRIMARY OUTCOMES:
The rate of H.pylori eradication | 4 weeks after finishing study drugs
  Helicobacter pylori eradication was assessed by ¹³C-urea breath test. [cutoff value(<4‰)]

SECONDARY OUTCOMES:
rate of drug compliance | 4 weeks after finishing study drugs
  good drug compliance measure by no of subjects taking >80% medicines
rate of side effects | 4 weeks after finishing study drugs
  Score side effects were mild, moderate or severe according to their influence on daily activities

CONTACTS AND LOCATIONS:
Overall Officials: I-Chen Wu, MD, PhD, Study Chair — Kaohsiung Medical University

IPD SHARING:
Plan to Share IPD: No